CLINICAL TRIAL: NCT02130843
Title: RETROSPECTIVE STUDY ABOUT A TECHNIQUE OF INSERTION OF TIEMANN MOUNTED URODYNAMIC CATHETER FOR DIFFICULT BLADDER CATHETERIZATION IN MALES
Brief Title: Tiemann Mounted Urodynamic Catheter Technique for Difficult Bladder Catheterization
Acronym: TMUC
Status: Completed | Type: Observational
Sponsor: Dr. Noam Kitrey (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Noam Kitrey, Urologist, Department of Urology, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Other Study IDs: SMC-13-0717
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: URINATION DISORDERS
Keywords: URINARY INCONTINENCE; URODYNAMICS; URINARY RETENTION; URINARY CATHETERIZATION
MeSH Terms: conditions — Urination Disorders; Urinary Incontinence; Urinary Retention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MALE PATIENTS BEFORE UDS: MALE PATIENTS BEFORE UDS WITH DIFFICULT CATHETERIZATION
  Interventions: Device: INSERTION OF URETEHRL CATHETER

INTERVENTIONS:
Device: INSERTION OF URETEHRL CATHETER — USE OF A TIEMANN CATHETER TO INSERT THE URODYNAMIC STUDY CATHETER INTO THE BLADDER
  Other Names: TIEMANN CATHETER

SUMMARY:
A report of a technique for insertion a soft urodynamic catheter into the bladder, when urethral obstruction causes the catheter to bend and fold over itself at the resistance site.

DETAILED DESCRIPTION:
The urodynamic catheter is mounted on a 12F Coudé tip Tiemann catheter, which then carries the tip of the urodynamic catheter beyond the obstruction site into the bladder.

The Tiemann catheter-mounted urodynamic catheter technique can serve as a suitable option to insert a urodynamic catheter into the bladder in all male patients in whom it fails due to kinking.

ELIGIBILITY:
Inclusion Criteria:

- MEN THAT UNDERWENT URODYNAMIC STUDY EVALUATION BETWEEN 6/2011 TO 9/2013

Exclusion Criteria:

NONE

-

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MALE PATIENTS 18-80 Y/O WHO UNDERWENT URODYNAMIC STUDY, AND HAD DIFFICULT CATHETERIZATION
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Successful Catheterization | Immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, IL, Israel